CLINICAL TRIAL: NCT04360473
Title: Ketamine Versus Magnesium Sulfate in the Time and Awakening Quality of General Anesthesia. Randomized Clinical Study.
Brief Title: Ketamine Versus Magnesium Sulfate in the Time and Awakening Quality of General Anesthesia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Associate professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE 28762619.0.0000.5448
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Awakening, Post-Anesthesia Delayed
Keywords: postoperative awakening; general anesthesia; magnesium sulfate; ketamine
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Anesthesia, General; Control Groups; Ketamine; Magnesium Sulfate; Magnesium

STUDY DESIGN:
Intervention Model Description: This is a prospective, controlled, covered and randomly distributed trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The person responsible for generating the sequence will use the result of the lottery to number the opaque envelopes and place the intervention corresponding to the group to which that lottery number belongs. This professional will not administer anesthesia to the patients in the study and will not participate in the collection or evaluation of the studied variables.
  The envelopes will be opened by professionals who will prepare the corresponding solution, keeping this information covered for the other members of the team and for the patients.
  The groups will be covered up for patients and for professionals who carry out the assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Active Comparator): The patients in this group will receive general balanced anesthesia
  Interventions: Other: General anesthesia
- Ketamine group (Experimental): The patients in this group will receive 0.3 mg / kg of ketamine in saline (total volume of 100 ml) 15 min before general balanced anesthetic induction
  Interventions: Drug: Ketamine plus general anesthesia
- Magnesium sulfate group (Experimental): The patients in this group will receive 40 mg / kg of magnesium sulfate in saline solution (total volume of 100 ml) 15 min before general balanced anesthetic induction
  Interventions: Drug: Magnesium sulfate plus general anesthesia
- Magnesium / ketamine group (Experimental): The patients in this group will receive 0.15 mg / kg of ketamine + 20 mg / kg of magnesium sulfate in saline solution (total volume of 100 ml) 15 min before general balanced anesthetic induction
  Interventions: Drug: ketamine plus magnesium sulfate plus general anesthesia

INTERVENTIONS:
Other: General anesthesia — Balanced general anesthesia. Induction with lidocaine, fentanyl, propofol and cisatracurium. Maintenance with sevoflurane.
  Other Names: Control group
  Arms: Control group
Drug: Ketamine plus general anesthesia — ketamine 0.3 mg / kg 15 minutes before balanced general anesthesia. Induction with lidocaine, fentanyl, propofol and cisatracurium. Maintenance with sevoflurane.
  Other Names: Ketamine group
  Arms: Ketamine group
Drug: Magnesium sulfate plus general anesthesia — Magnesium sulfate 40 mg / kg 15 minutes before balanced general anesthesia. Induction with lidocaine, fentanyl, propofol and cisatracurium. Maintenance with sevoflurane.
  Other Names: Magnesium sulfate group
  Arms: Magnesium sulfate group
Drug: ketamine plus magnesium sulfate plus general anesthesia — Ketamine 0.15 mg/kg plus magnesium sulfate 20 mg/kg 15 minutes before balanced general anesthesia. Induction with lidocaine, fentanyl, propofol and cisatracurium. Maintenance with sevoflurane
  Other Names: Magnesium / ketamine group
  Arms: Magnesium / ketamine group

SUMMARY:
The introduction of the laparoscopic technique for cholecystectomy significantly reduced the incidence and intensity of postoperative pain, with improvement in other markers, such as patient satisfaction, and reduction in hospital stay. However, pain in the postoperative period of laparoscopic cholecystectomy is still a concern that challenges modern anesthesiology. Ketamine and magnesium sulfate are two blockers of N-methyl-D-aspartate (NMDA) receptors with the ability to reduce postoperative pain and postoperative opioid consumption. A frequent concern among anesthesiologists is the quality and time of awakening in patients receiving these medications The main objective of this trial is to compare the quality and time of awakening in patients receiving magnesium sulfate or ketamine.

The secondary objective is to compare postoperative analgesia during the postoperative hospital stay.

Hypothesis: Our hypothesis is that patients have a faster awakening when they receive magnesium sulfate as an analgesic adjunct, when compared to patients who receive ketamine .

Design: this is a prospective, controlled, covered and randomly distributed trial.

DETAILED DESCRIPTION:
Intervention: the sample of participants will be distributed in 4 groups. The placebo (PG) group will receive 100 ml of saline solution 15 min before anesthetic induction. The ketamine group (KG) will receive 0.3 mg / kg of ketamine in saline (total volume of 100 ml) 15 min before anesthetic induction. The magnesium sulfate group (SG) will receive 40 mg / kg of magnesium sulfate in saline solution (total volume of 100 ml) 15 min before anesthetic induction. The mixed group (MG) will receive 0.15 mg / kg of ketamine + 20 mg / kg of magnesium sulfate in saline solution (total volume of 100 ml) 15 min before anesthetic induction. All participants will be submitted to balanced anesthesia. Anesthetic induction will be started after 5 min of pre-oxygenation, with lidocaine 1.5 mg / kg, fentanyl 3 µg / kg, propofol until clinical hypnosis, cisatracurium 0.1 mg / kg and intubation after adequate neuromuscular relaxation. Maintenance will be with sevoflurane in concentration under clinical demand, repeating boluses of fentanyl 1 µg / kg and cisatracurium 0.03 mg / kg, as needed.

Primary Outcomes: time between the end of anesthetic administration and bispectral index (BIS) > 60, and a battery of neuropsychological tests to assess postoperative cognitive dysfunction tested in the Brazilian population 3 h after the end of anesthetic administration.

Secondary Outcomes: response to the brief pain inventory questionnaire and opioid consumption in the first 2 postoperative days.

Recruitment and timeline : patients will be recruited in the pre-anesthetic evaluation and assessments will be made of covertly in the immediate postoperative period and during the two days after surgery, being registered the pain scores and the consumption of opioids.

Sample calculation: the sample of 120 participants was calculated with a 95% confidence index and 80% statistical power. To compensate for losses, 140 individuals will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo laparoscopic cholecystectomy, agreement to voluntarily participate in the trial and sign the free and informed consent form.

Exclusion Criteria:

* Coronary disease, ventricular atrial block II or worse, with renal failure , previous history of brain disease, dementia or other psychiatric diseases, and patients with a body mass index> 35 kg / m² , allergy to any products used in the trial, preoperative use of opioids or corticosteroids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time for awakening | Three hours
  Time, after the end of anesthetic administration, to get the bispectral index (BIS) > 60.
Awakening quality | Three hours
  Questions related to name, place, time, reason for hospitalization and verbal learning test, consisting of 15 words that the patient will be asked to repeat 20 minutes after hearing them. The wrong answers will be compared among groups.

SECONDARY OUTCOMES:
Postoperative pain | Two days
  Verbal pain score 0 (without pain) to 10 (worst imaginable pain), and the effect of pain over humor, ambulation and sleep, each one 0 (without effect) to 10 (worst imaginable effect)
Postoperative analgesia | Two days
  Opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Vieira, Principal Investigator — University of Sao Paulo School of Medicine
Locations (1):
- Hospital da Beneficência Portuguesa de Santos, Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] REFERENCES 1. Hendolin HI, Pääkkönen ME, Alhava EM, Tarvainen R, Kemppinen T, Lahtinen. Laparoscopic or open cholecystectomy: a prospective randomized trial to compare postoperative pain, pulmonary function, and stress response. Eur J Surg. 2000; 166: 394-9. 2. Attwood SEA, Hill ADK, Mealy K, Stephens RB. A prospective comparison of laparoscopic versus open cholecystectomy. Annlas of the Royal College of Surgeons of England. 1992; 74: 397-400. 3. Keus F, by Jong J, Gooszen HG, Laarhoven CJHM. Laparoscopic versus open cholecystectomy for patients with symptomatic cholecystolithiasis. Cochrane Database of Systematic Reviews. 2006, Issue 4. Art. No.: CD006231. 4. Barazanchi AWH, MacFater WS, Rahiri JL, Tutone S, Hill AG, Joshi GP. Evidence-based management of pain after laparoscopic cholecystectomy: a PROSPECT review update. Br J Anaesth. 2018; 121: 787-803. 5. Bisgaard T, Klarskov B, Rosenberg J, Kehlet H. Characteristics and prediction of early pain after laparoscopic cholecystectomy. Pain. 2001 ; 90: 261-9. 6. Ye Fan, Wu Y, Zhou C. Effect of intravenous ketamine for postoperative analgesia in patients undergoing laparoscopic cholecystectomy. Meta-analysis. Medicine. 2017; 96: 51 7. Launo C, Bassi C, Spagnolo L, Badano S, Ricci C, Lizzi A, et al. Preemptive ketamine during general anesthesia for postoperative analgesia in patients undergoing laparoscopic cholecystectomy. Minerva Anestesiol. 2004; 70: 727-38. 8. Hang LH, Shao DH, Gu YP. The ED50 and ED95 of ketamine for prevention of postoperative hyperalgesia after remifentanil-based anesthesia in patients undergoing laparoscopic cholecystectomy. Swiss Med Wkly. 2011; 141: w13195 . 9. Minds O, Harlak A, Yigit T, Balkan A, Balkan M, Cosar A, et al. Effect of intraoperative magnesium sulphate infusion on pain relief after laparoscopic cholecystectomy. Acta Anaesthesiol Scand. 2008; 52: 1353-9. 10. Chen C, Tao R. The impact of magnesium sulfate on pain control after laparoscopic cholecystectomy: a meta-analysis of randomized controlled studies. Surg Laparosc Endosc Percutan. 2018; 28: 349-53. 11. Valentin LSS, Pietrobon R, Junior WA, et al. Definition and application of a battery of neuropsychological tests to assess postoperative cognitive dysfunction. Einstein. 2015; 13: 20-6.